CLINICAL TRIAL: NCT06202027
Title: Post Marketing Surveillance Study to Observe Safety and Effectiveness of CRYSVITA® in S. Korean Patients
Status: Recruiting | Type: Observational
Sponsor: Kyowa Kirin Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: CRYSVITA PMS
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: FGF23-related Hypophosphataemic Rickets and Osteomalacia
MeSH Terms: conditions — Osteomalacia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: FGF23-related hypophosphataemic rickets and osteomalacia — FGF23-related hypophosphataemic rickets and osteomalacia

SUMMARY:
The objective of this post-marketing surveillance (PMS) study is to assess the safety and effectiveness of CRYSVITA injection 10, 20, and 30mg, equivalent to in routine clinical settings

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been started on CRYSVITA® in accordance with the approved label in Korea
2. Those (or his/her legal guardian) who have agreed in writing to participate in the survey. Children who have obtained a written consent of his/her legal guardian about participation in this survey. In case of pediatric patient, explain sufficiently what you think the patient can understand. In this case, the legal guardian may provide supplementary explanations of the survey.

Exclusion Criteria:

1. Patients for whom Burosumab is contraindicated according local label of CRYSVITA®
2. Patients who intend to use this drug for other purposes
3. Patients who participated in pre-market clinical trials with CRYSVITA® (Consecutive investigation method ONLY)
4. Patients who have been taking this drug before the starting day of this study (Consecutive investigation method ONLY)

Min Age: 1 Day | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: FGF23-related hypophosphataemic rickets and osteomalacia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2031-06-16 (Estimated); Study Completion 2031-07-16 (Estimated)

PRIMARY OUTCOMES:
safety (Special situation, adverse event, symptom, or disease occuring during treatment with a drug) | 4 weeks after follow up
  Investigators have to record all events (i.e., all AEs and special situations) in CRFs including undesirable medical findings obtained during the medical examination as well as spontaneous reports from subjects. All AEs occurring for at least 4 weeks after the last dose of CRYSVITA® should be included in this study

SECONDARY OUTCOMES:
Serum Phosphorus Concentration | 24 weeks
  1) Change from baseline over time in Serum Phosphorus Concentration (mg/dL), up to Week 24
1,25-Dihydroxyvitamin D | 24 weeks
  2) Change from baseline over time in 1,25-Dihydroxyvitamin D, up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: HaeMi Park, Study Director — Kyowa Kirin Korea Co., Ltd.
Locations (10):
- South Korea (10):
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Yangsan Pusan National University Hospital, Yangsan, Gyeongsangnam-do
  - Chonnam National University Hospital, Gwangju, Jeollanam-do
  - Chungnam National University Sejong Hospital, Sejong, Sejong Special Self-Governing City
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
Undecided